CLINICAL TRIAL: NCT00410761
Title: An International, Phase III, Randomized, Double-Blinded, Placebo-Controlled, Multi-Center Study to Assess the Efficacy of ZD6474 (ZACTIMATM) Versus Placebo in Subjects With Unresectable Locally Advanced or Metastatic Medullary Thyroid Cancer
Brief Title: An Efficacy Study Comparing ZD6474 to Placebo in Medullary Thyroid Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4200C00058; LPS14811 (Other: Sanofi Identifier); 2005-005077-29 (EudraCT Number)
Record Dates: First submitted 2006-12-06; First posted 2006-12-13 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Cancer
Keywords: ZD6474; MTC; Hereditary Medullary Thyroid Cancer; Sporadic Medullary Thyroid Cancer; Medullary Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms; Familial medullary thyroid carcinoma; Carcinoma, Medullary | interventions — vandetanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (No Intervention): Placebo vandetanib
- 2 (Experimental): Vandetanib
  Interventions: Drug: ZD6474 (Vandetanib)

INTERVENTIONS:
Drug: ZD6474 (Vandetanib) — once daily oral tablet
  Other Names: ZACTIMA™; SAR390530
  Arms: 2

SUMMARY:
The purpose of this study is to learn how hereditary or sporadic medullary thyroid cancer patients, treated with ZD6474, react to the drug, what happens to ZD6474 in the human body, about the side effects of ZD6474, and if ZD6474 can decrease or prevent the growth of tumors.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of unresectable, locally advanced or metastatic hereditary or sporadic Medullary Thyroid Cancer.
* Presence of measurable tumor
* Able to swallow medication

Exclusion Criteria:

* Major surgery within 4 weeks before randomization
* Last dose of prior chemotherapy received less than 4 weeks prior to randomization
* Radiation therapy within the last 4 weeks prior to randomization(with exception of palliative radiotherapy)
* Brain metastases or spinal cord compression, unless treated at least 4 weeks before first dose and stable without steroid treatment for 10 days
* Significant cardiac events
* Previous ZD6474 treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2006-11-23 (Actual); Primary Completion 2009-07-31 (Actual); Study Completion 2024-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (127):
- United States (32):
  - Investigational Site Number 3, Little Rock, Arkansas
  - University Arkansas Site Number : 3, Little Rock, Arkansas
  - Investigational Site Number 8, San Francisco, California
  - USCF / Mt Zion Medical Center Site Number : 8, San Francisco, California
  - Investigational Site Number 9, Aurora, Colorado
  - University Of Colorado Health Sciences Center Site Number : 9, Aurora, Colorado
  - Investigational Site Number 11, New Haven, Connecticut
  - Yale University School Medicine Site Number : 11, New Haven, Connecticut
  - Investigational Site Number 15, Jacksonville, Florida
  - Mayo Clinic- Site Number : 15, Jacksonville, Florida
  - Investigational Site Number 18, Chicago, Illinois
  - The University Of Chicago Site Number : 18, Chicago, Illinois
  - Investigational Site Number 17, Lexington, Kentucky
  - The University Of Kentucky Site Number : 17, Lexington, Kentucky
  - Dana Farber Cancer Institute Site Number : 2, Boston, Massachusetts
  - Investigational Site Number 2, Boston, Massachusetts
  - Investigational Site Number 7, Detroit, Michigan
  - Wayne State University / Harper Hospital Site Number : 7, Detroit, Michigan
  - Investigational Site Number 14, Rochester, Minnesota
  - Mayo Clinic- Site Number : 14, Rochester, Minnesota
  - Investigational Site Number 10, St Louis, Missouri
  - Washington University School Of Med Site Number : 10, St Louis, Missouri
  - Investigational Site Number 6, Cincinnati, Ohio
  - University Of Cincinnati Site Number : 6, Cincinnati, Ohio
  - Investigational Site Number 22, Portland, Oregon
  - Oregon Health & Science University- Site Number : 22, Portland, Oregon
  - Investigational Site Number 19, Charleston, South Carolina
  - Medical University of South Carolina- Site Number : 19, Charleston, South Carolina
  - Anderson Cancer Center Site Number : 13, Houston, Texas
  - Investigational Site Number 13, Houston, Texas
  - Fletcher Allen Health Care Site Number : 21, Burlington, Vermont
  - Investigational Site Number 21, Burlington, Vermont
- Investigational Site Number 1001, St Leonards, Australia
- Austria (2):
  - Investigational Site Number 1901, Vienna
  - Investigational Site Number : 1901, Vienna
- Belgium (4):
  - Investigational Site Number : 1101, Anderlecht
  - Investigational Site Number 1101, Brussels
  - Investigational Site Number 1102, Leuven
  - Investigational Site Number : 1102, Leuven
- Brazil (4):
  - Hospital De Clinicas De Porto Alegre- Site Number : 2301, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina de Ribeirao Preto - USP- Site Number : 2302, Ribeirão Preto, São Paulo
  - Investigational Site Number 2301, Porto Alegre
  - Investigational Site Number 2302, Ribeirão Preto
- Canada (10):
  - Investigational Site Number : 1203, Calgary, Alberta
  - Investigational Site Number : 1201, Moncton, New Brunswick
  - Investigational Site Number : 1202, London, Ontario
  - Investigational Site Number : 1205, Toronto, Ontario
  - Investigational Site Number : 1204, Sherbrooke, Quebec
  - Investigational Site Number 1203, Calgary
  - Investigational Site Number 1202, London
  - Investigational Site Number 1201, Moncton
  - Investigational Site Number 1204, Sherbrooke
  - Investigational Site Number 1205, Toronto
- Czechia (2):
  - Investigational Site Number 3601, Prague
  - Investigational Site Number : 3601, Prague
- Denmark (2):
  - Investigational Site Number 2701, Odense C
  - Investigational Site Number : 2701, Odense C
- France (6):
  - Investigational Site Number 2802, Bordeaux
  - Investigational Site Number : 2802, Bordeaux
  - Investigational Site Number 2803, Lyon
  - Investigational Site Number : 2803, Lyon
  - Investigational Site Number 2801, Villejuif
  - Investigational Site Number : 2801, Villejuif
- Germany (6):
  - Investigational Site Number 2002, Essen
  - Investigational Site Number : 2002, Essen
  - Investigational Site Number 2001, Halle
  - Investigational Site Number : 2001, Halle
  - Investigational Site Number 2005, Würzburg
  - Investigational Site Number : 2005, Würzburg
- Hungary (2):
  - Investigational Site Number 1601, Pécs
  - Investigational Site Number : 1601, Pécs
- India (4):
  - Investigational Site Number 1401, Mumbai
  - Investigational Site Number : 1401, Mumbai
  - Investigational Site Number 1402, Vellore
  - Investigational Site Number : 1402, Vellore
- Italy (12):
  - Investigational Site Number 2506, Catania
  - Investigational Site Number : 2506, Catania
  - Investigational Site Number 2502, Milan
  - Investigational Site Number : 2502, Milan
  - Investigational Site Number 2503, Napoli
  - Investigational Site Number : 2503, Napoli
  - Investigational Site Number 2501, Pisa
  - Investigational Site Number : 2501, Pisa
  - Investigational Site Number 2505, Roma
  - Investigational Site Number : 2505, Roma
  - Investigational Site Number 2504, Siena
  - Investigational Site Number : 2504, Siena
- Mexico (4):
  - Investigational Site Number 2403, Ciudad Madero
  - Investigational Site Number 2402, Mexico City
  - Investigational Site Number 2404, México
  - Investigational Site Number : 2404, México
- Netherlands (4):
  - Investigational Site Number 2902, Groningen
  - Investigational Site Number : 2902, Groningen
  - Investigational Site Number 2901, Utrecht
  - Investigational Site Number : 2901, Utrecht
- Poland (6):
  - Investigational Site Number : 1702, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 1703, Warsaw, Masovian Voivodeship
  - Investigational Site Number 1701, Gliwice
  - Investigational Site Number : 1701, Gliwice
  - Investigational Site Number 1702, Poznan
  - Investigational Site Number 1703, Warsaw
- Portugal (3):
  - Investigational Site Number 2602, Coimbra
  - Investigational Site Number 2601, Lisbon
  - Investigational Site Number : 2601, Lisbon
- Investigational Site Number 1801, Bucharest, Romania
- Russia (2):
  - Investigational Site Number 3301, Obninsk
  - Investigational Site Number : 3301, Obninsk
- Serbia (4):
  - Investigational Site Number 3401, Belgrade
  - Investigational Site Number : 3401, Belgrade
  - Investigational Site Number 3402, Belgrade
  - Investigational Site Number : 3402, Belgrade
- South Korea (2):
  - Investigational Site Number : 1501, Seoul
  - Investigational Site Number 1501, Seoul
- Spain (6):
  - Investigational Site Number : 3002, Pamplona, Navarre
  - Investigational Site Number 3003, Madrid
  - Investigational Site Number : 3003, Madrid
  - Investigational Site Number 3001, Madrid
  - Investigational Site Number : 3001, Madrid
  - Investigational Site Number 3002, Pamplona
- Sweden (4):
  - Investigational Site Number 3102, Stockholm
  - Investigational Site Number : 3102, Stockholm
  - Investigational Site Number 3101, Uppsala
  - Investigational Site Number : 3101, Uppsala
- Switzerland (4):
  - Investigational Site Number 2101, Basel
  - Investigational Site Number : 2101, Basel
  - Investigational Site Number 2102, Bern
  - Investigational Site Number : 2102, Bern

REFERENCES:
- [Result] Wells SA Jr, Robinson BG, Gagel RF, Dralle H, Fagin JA, Santoro M, Baudin E, Elisei R, Jarzab B, Vasselli JR, Read J, Langmuir P, Ryan AJ, Schlumberger MJ. Vandetanib in patients with locally advanced or metastatic medullary thyroid cancer: a randomized, double-blind phase III trial. J Clin Oncol. 2012 Jan 10;30(2):134-41. doi: 10.1200/JCO.2011.35.5040. Epub 2011 Oct 24. PMID 22025146
- See also: CSR-D4200C00058.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=348&filename=CSR-D4200C00058.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 331 participants were enrolled in the study. The study was conducted at 60 study sites in 23 countries. First participant enrolled 23 November 2006, last participant enrolled 19 October 2007.
Groups:
- Vandetanib 300 mg/Vandetanib 300 mg: Participants received vandetanib 300 mg orally once daily until objective disease progression, any other withdrawal criteria was met or at the investigator's discretion, the approval and implementation of protocol amendment 6 during the blinded randomized treatment period. Upon disease progression or implementation of protocol amendment 6, participants who were unblinded were given the option to enter the open-label treatment period and continue to receive vandetanib 300 mg orally once daily for as long as they still benefitted of it per investigator judgement or until they were given another anti-cancer therapy.
- Placebo/Vandetanib 300 mg: Participants received placebo matched to vandetanib orally once daily until objective disease progression, any other withdrawal criteria was met or at the investigator's discretion, the approval and implementation of protocol amendment 6 during the blinded randomized treatment period. Upon disease progression or implementation of protocol amendment 6, participants who were unblinded were given the option to enter the open-label treatment period and receive vandetanib 300 mg orally once daily for as long as they still benefitted of it per investigator judgement or until they were given another anti-cancer therapy.
Period: Randomized Treatment Period
Arm/Group | Vandetanib 300 mg/Vandetanib 300 mg | Placebo/Vandetanib 300 mg
Started (Randomized participants.) | 231 | 100
Received Randomized Treatment | 231 | 99
Completed (Participants who ended randomized treatment.) | 14 | 1
Not Completed | 217 | 99
Not completed — Adverse Event | 34 | 3
Not completed — Objective Disease Progression | 103 | 68
Not completed — Withdrawal by Subject | 11 | 6
Not completed — Other | 69 | 21
Not completed — Randomized but did not Receive Treatment | 0 | 1
Period: Open-Label Treatment Period
Arm/Group | Vandetanib 300 mg/Vandetanib 300 mg | Placebo/Vandetanib 300 mg
Started (Participants who discontinued randomized treatment and received open-label treatment (vandetanib 300 mg).) | 109 | 79
Completed (Participants who ended open-label treatment (vandetanib 300 mg).) | 28 | 21
Not Completed | 81 | 58
Not completed — Adverse Event | 13 | 15
Not completed — Objective Disease Progression | 42 | 27
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Other | 18 | 9

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants.
Groups:
- Vandetanib 300 mg: Vandetanib (300 mg daily)
- Placebo: Placebo daily
- Total: Total of all reporting groups
Arm/Group | Vandetanib 300 mg | Placebo | Total
Number analyzed (Participants) | 231 | 100 | 331
Age, Continuous [Mean (Full Range); unit: years] | 50.7 [18 to 83] | 53.4 [26 to 84] | 52 [18 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 44 | 141
  Male | 134 | 56 | 190

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival(PFS)
Description: Median time to progression (months) from randomisation until objective disease progression (determined by RECIST assessments) or death (by any cause in the absence of objective progression) provided death is within 3 months from the last evaluable RECIST assessment. Values here are estimated (from a Weibull model) as the medians were not met.
Time Frame: RECIST tumour assessments were performed at screening (within 3 weeks before date of randomisation), then once every 12 weeks up to and including discontinuation of blinded study treatment, unless patients had withdrawn consent.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 231 | 100
Months | 30.5 [NA to NA] — PFS is a time to event endpoint and because the medians were not met in this study there is no appropriate measure of dispersion of the median | 19.2 [NA to NA] — PFS is a time to event endpoint and because the medians were not met in this study there is no appropriate measure of dispersion of the median

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is the number of patients that are responders ie those patients with a confirmed best objective response of complete response (CR) or partial response (PR) as defined by RECIST criteria.
  The categories for best objective response are CR, PR, stable disease (SD)>= 12 weeks, progressive disease (PD) or NE.
Time Frame: RECIST assessments performed at screening (within 3 weeks before randomisation), then every 12 weeks. For patients with objective response of CR or PR, an additional confirmatory scan was performed ≥4 weeks following the date of first response.
Measure: Number; unit: Participants
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 231 | 100
Participants | 104 | 13

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate is defined as the number of patients who achieved disease control at 8 weeks following randomisation. Disease control at 8 weeks is defined as a best objective response of complete response (CR), partial response (PR) or stable disease (SD) >= 12 weeks
Time Frame: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 231 | 100
Participants | 200 | 71

4. Secondary Outcome: Duration of Response (DoR)
Description: Response is defined as a confirmed best objective response of CR or PR. Duration of response is defined as time from the date of first documented response until date of documented progression or death in the absence of disease progression (provided death is within 3 months of last RECIST assessment). Values are estimated as the medians weren't met
Time Frame: as for outcome 1
Population: DoR is a time to event endpoint and because the medians were not met in this study there is no appropriate measure of dispersion of the median
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 104 | 13
Months | 22.2 [NA to NA] — DoR is a time to event endpoint and because the medians were not met in this study there is no appropriate measure of dispersion of the median | 16.3 [NA to NA] — DoR is a time to event endpoint and because the medians were not met in this study there is no appropriate measure of dispersion of the median

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization until death.
Time Frame: From date of randomization until death, up to approximately 105 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 231 | 100
Months | 81.6 [64.6 to 98.5] | 80.4 [52.5 to NA] — NA indicates that the upper limit of confidence interval was not estimable due to insufficient number of participants with events.

6. Secondary Outcome: Biochemical Response Calcitonin (CTN)
Description: Best biochemical response was calculated from assessments at baseline and during treatment. Responders were those patients with a best biochemical response of CR or PR, confirmed by repeat assessments, which were to be performed no less than 4 weeks after the criteria for PR or CR were first met. CR and PR being defined according to level of CTN.
Time Frame: Blood samples for analysis of CTN were taken at screening baseline (average of 0, 1, 4 and 8 hours), then every 4 weeks until discontinuation and 60 day follow up
Measure: Number; unit: Participants
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 231 | 100
Participants | 160 | 3

7. Secondary Outcome: Biochemical Response Carcinoembryonic Antigen (CEA)
Description: Best biochemical response was calculated from assessments at baseline and during treatment. Responders were those patients with a best biochemical response of CR or PR, confirmed by repeat assessments, which were to be performed no less than 4 weeks after the criteria for PR or CR were first met. CR and PR being defined according to level of CEA.
Time Frame: Blood samples for analysis of CEA were taken at screening baseline (average of 0, 1, 4 and 8 hours), then every 4 weeks until discontinuation and 60 day follow up
Measure: Number; unit: Participants
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 231 | 100
Participants | 119 | 2

8. Secondary Outcome: Time to Worsening of Pain (TWP)
Description: TWP was derived using the worst pain score from brief pain inventory (BPI) and patient reported opioid analgesic use. BPI uses 0 to 10 numeric rating scales asking subjects to rate their pain. TWP results are presented.
Time Frame: During the last week of the screening period (Day -7 to Day 0), the brief pain inventory (BPI) and opioid analgesic use were self-reported once a day for 4 days to establish baseline, then every week during blinded study treatment, up to discontinuation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 231 | 100
Months | 7.85 [5.39 to 12.16] | 3.25 [1.87 to 5.26]

ADVERSE EVENTS:
Time Frame: Serious adverse events(SAEs) and all-cause mortality(deaths) were collected from randomization (Day 1) up to end of follow-up, approximately 212 months. Other (non-serious) AEs were reported from randomization (Day 1) up to data cut-off date 01-Jun-2010, approximately 42 months. AEs and SAEs were collected from Day 1 to cut-off date 01-Jun-2010 and were presented in clinical database. After this cut-off date, SAEs were reported in pharmacovigilance database, but no non-serious AEs were reported.
Description: The safety population included all participants who received at least 1 dose of vandetanib/placebo. All-cause mortality (deaths) was assessed in all randomized participants.
Groups:
- Randomized Treatment Period: Vandetanib 300 mg: Participants received vandetanib 300 mg orally once daily until objective disease progression, any other withdrawal criteria was met or at the investigator's discretion, the approval and implementation of protocol amendment 6 during the blinded randomized treatment period.
- Randomized Treatment Period: Placebo: Participants received placebo matched to vandetanib orally once daily until objective disease progression, any other withdrawal criteria was met or at the investigator's discretion, the approval and implementation of protocol amendment 6 during the blinded randomized treatment period.
- Open-Label Treatment Period: Vandetanib 300 mg/Vandetanib 300 mg: Participants who received vandetanib 300 mg during the blinded randomized treatment period and who were unblinded due to disease progression or as a result of protocol amendment 6 were given the option to continue to receive vandetanib 300 mg orally once daily in the open-label treatment period for as long as they still benefitted of it per investigator judgement or until they were given another anti-cancer therapy.
- Open-Label Treatment Period: Placebo/Vandetanib 300 mg: Participants who received placebo matched to vandetanib during the blinded randomized treatment period and who were unblinded due to disease progression or as a result of protocol amendment 6 were given the option to receive vandetanib 300 mg orally once daily in the open-label treatment period for as long as they still benefitted of it per investigator judgement or until they were given another anti-cancer therapy.
Arm/Group | Randomized Treatment Period: Vandetanib 300 mg | Randomized Treatment Period: Placebo | Open-Label Treatment Period: Vandetanib 300 mg/Vandetanib 300 mg | Open-Label Treatment Period: Placebo/Vandetanib 300 mg
All-Cause Mortality (participants affected / at risk) | 66/231 | 10/100 | 52/109 | 41/79
Serious Adverse Events (participants affected / at risk) | 92/231 | 16/99 | 53/109 | 36/79
Other Adverse Events (participants affected / at risk) | 226/231 | 87/99 | 32/109 | 70/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Treatment Period: Vandetanib 300 mg (N=231) | Randomized Treatment Period: Placebo (N=99) | Open-Label Treatment Period: Vandetanib 300 mg/Vandetanib 300 mg (N=109) | Open-Label Treatment Period: Placebo/Vandetanib 300 mg (N=79)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular Insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial Haemorrhage (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Patent Ductus Arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cushing's Syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal Artery Occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 0 (0) | 1 (2) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mechanical Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Obstructive Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pancreatitis Chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumatosis Intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reflux Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Asthenia (General disorders) | 2 (3) | 0 (0) | 1 (2) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Device Occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
General Physical Health Deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sudden Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iodine Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal Wall Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 2 (2)
Appendicitis Perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bartholin's Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bronchitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Gastroenteritis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected Bites (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peridiverticular Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (9) | 0 (0) | 3 (5) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (4) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcal Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 3 (6) | 0 (0) | 2 (2) | 0 (0)
Urinary Tract Infection Pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exposure During Pregnancy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaw Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Haematuria (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venomous Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound Necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-Reactive Protein Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International Normalised Ratio Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic Specific Antigen Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (9)
Breast Cancer Female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colorectal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Germ Cell Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular Seminoma (Pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain Oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cerebellar Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral Ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depressed Level Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Internal Capsule Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Subarachnoid Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bipolar Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Completed Suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus Ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (4) | 0 (0) | 0 (0) | 3 (3)
Obstructive Uropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual Bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Accelerated Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jugular Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic Venous Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vena Cava Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Treatment Period: Vandetanib 300 mg (N=231) | Randomized Treatment Period: Placebo (N=99) | Open-Label Treatment Period: Vandetanib 300 mg/Vandetanib 300 mg (N=109) | Open-Label Treatment Period: Placebo/Vandetanib 300 mg (N=79)
Vertigo (Ear and labyrinth disorders) | 10 (12) | 2 (2) | 1 (1) | 5 (5)
Hypothyroidism (Endocrine disorders) | 16 (19) | 0 (0) | 1 (1) | 1 (1)
Corneal Opacity (Eye disorders) | 11 (11) | 0 (0) | 0 (0) | 4 (4)
Vision Blurred (Eye disorders) | 19 (23) | 1 (1) | 1 (1) | 5 (5)
Abdominal Pain (Gastrointestinal disorders) | 33 (50) | 5 (6) | 2 (2) | 5 (6)
Abdominal Pain Upper (Gastrointestinal disorders) | 23 (33) | 7 (7) | 1 (1) | 5 (5)
Constipation (Gastrointestinal disorders) | 14 (21) | 5 (5) | 3 (3) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 123 (180) | 27 (36) | 4 (5) | 32 (39)
Dry Mouth (Gastrointestinal disorders) | 22 (22) | 3 (3) | 0 (0) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 28 (33) | 4 (5) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 74 (97) | 16 (16) | 5 (5) | 18 (24)
Toothache (Gastrointestinal disorders) | 7 (7) | 5 (17) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 33 (45) | 7 (7) | 3 (5) | 9 (9)
Asthenia (General disorders) | 34 (39) | 12 (12) | 0 (0) | 12 (13)
Fatigue (General disorders) | 54 (64) | 23 (27) | 3 (3) | 13 (16)
Pyrexia (General disorders) | 18 (20) | 3 (3) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 11 (11) | 6 (8) | 0 (0) | 2 (2)
Folliculitis (Infections and infestations) | 8 (9) | 1 (1) | 0 (0) | 5 (5)
Influenza (Infections and infestations) | 16 (16) | 3 (3) | 2 (2) | 3 (4)
Nasopharyngitis (Infections and infestations) | 29 (43) | 9 (12) | 2 (4) | 4 (6)
Upper Respiratory Tract Infection (Infections and infestations) | 19 (27) | 3 (5) | 2 (2) | 8 (13)
Urinary Tract Infection (Infections and infestations) | 16 (27) | 6 (7) | 1 (3) | 5 (6)
Electrocardiogram Qt Prolonged (Investigations) | 32 (46) | 1 (1) | 3 (3) | 7 (8)
Weight Decreased (Investigations) | 27 (28) | 10 (10) | 2 (2) | 5 (5)
Weight Increased (Investigations) | 6 (6) | 0 (0) | 0 (0) | 4 (4)
Decreased Appetite (Metabolism and nutrition disorders) | 42 (53) | 13 (13) | 2 (3) | 17 (19)
Hypocalcaemia (Metabolism and nutrition disorders) | 22 (27) | 3 (4) | 3 (3) | 7 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (24) | 10 (13) | 2 (2) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 23 (37) | 20 (41) | 6 (9) | 3 (3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 5 (5) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 14 (16) | 1 (2) | 0 (0) | 4 (5)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 18 (24) | 6 (7) | 2 (2) | 2 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 12 (20) | 10 (14) | 3 (3) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 2 (2) | 2 (2) | 4 (4)
Neck Pain (Musculoskeletal and connective tissue disorders) | 17 (20) | 9 (10) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 17 (24) | 14 (17) | 3 (3) | 6 (6)
Dizziness (Nervous system disorders) | 21 (24) | 5 (5) | 1 (1) | 7 (7)
Dysgeusia (Nervous system disorders) | 20 (22) | 3 (3) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 62 (138) | 9 (13) | 4 (6) | 5 (5)
Paraesthesia (Nervous system disorders) | 13 (15) | 3 (3) | 2 (4) | 4 (5)
Tremor (Nervous system disorders) | 7 (7) | 0 (0) | 1 (1) | 4 (4)
Anxiety (Psychiatric disorders) | 12 (13) | 5 (5) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 22 (25) | 3 (3) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 32 (36) | 12 (12) | 1 (1) | 6 (6)
Proteinuria (Renal and urinary disorders) | 23 (26) | 2 (3) | 1 (1) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (31) | 10 (15) | 3 (3) | 3 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 3 (3) | 1 (1) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 10 (14) | 3 (4) | 11 (11)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 5 (6) | 0 (0) | 3 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 0 (0) | 4 (4)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 20 (32) | 6 (14) | 1 (1) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 47 (66) | 5 (5) | 0 (0) | 21 (25)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (19) | 0 (0) | 2 (2) | 4 (4)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 35 (45) | 2 (4) | 0 (0) | 4 (6)
Dry Skin (Skin and subcutaneous tissue disorders) | 36 (41) | 5 (5) | 0 (0) | 11 (14)
Erythema (Skin and subcutaneous tissue disorders) | 22 (22) | 3 (3) | 0 (0) | 6 (8)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 29 (33) | 0 (0) | 0 (0) | 11 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 26 (31) | 4 (5) | 0 (0) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 105 (158) | 11 (12) | 4 (4) | 25 (40)
Hypertension (Vascular disorders) | 71 (79) | 6 (6) | 2 (2) | 15 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.